CLINICAL TRIAL: NCT05317442
Title: Open-label Study to Evaluate the Efficacy and Safety of Fespixon Cream for the Treatment of Pressure Injury in Sacrum and Greater Trochanter Wound
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume.
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hsian-Jenn Wang, Consultant, Department of Surgery, Taipei Medical University WanFang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ON101CLAS05
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Pressure Injury Stage 2
Keywords: Fespixon; Pressure Injury; Wound; NPIAP Stage 2
MeSH Terms: conditions — Pressure Ulcer; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: 1. Uncontrolled
  2. Open-label
  3. Randomized: N/A
  4. Single Arm
  5. Duration of treatment: up to 16 weeks
  6. Titration: no
  7. Multi-center(Taiwan)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pressure Injury in Sacrum and Greater Trochanter Wound (Experimental): 1. Name: Fespixon Cream
  2. Dosage form: Topical cream, 15 g ointment per tube
  3. Active ingredients: 1.25% extracts of Plectranthus amboinicus (PA-F4, 0.25%) and Centella asiatica (S1, 1%)
  4. Dose(s): Apply 1 cc per 5 cm^2 ulcer size (not exceeding 2 mm in thickness)
  5. Dosing schedule: Apply once a day
  6. Duration: up to 16 weeks
  Interventions: Drug: Fespixon Cream

INTERVENTIONS:
Drug: Fespixon Cream — 1. Name: Fespixon Cream
  2. Dosage form: Topical cream, 15 g ointment per tube
  3. Active ingredients: 1.25% extracts of Plectranthus amboinicus (PA-F4, 0.25%) and Centella asiatica (S1, 1%)
  4. Dose(s): Apply 1 cc per 5 cm^2 ulcer size (not exceeding 2 mm in thickness)
  5. Dosing schedule: Apply once a day
  6. Duration: up to 16 weeks
  Other Names: ON101 Cream

SUMMARY:
Open-label Study to Evaluate the Efficacy and Safety of Fespixon Cream for the Treatment of Pressure Injury in Sacrum and Greater Trochanter Wound

DETAILED DESCRIPTION:
This study is designed as a single-arm, open-label, multi-center study to evaluate the efficacy and safety of Fespixon Cream for the treatment of pressure injury in sacrum wound. The duration of this study is: run in/ screen phase (2 weeks); treatment phase (16 weeks); follow-up phase (4 weeks), and visits are conducted every 2 weeks for a total of 12 visits. During the treatment phase, the Fespixon cream will be applied to the target ulcer once a day for a maximum period of 16 weeks, until the wound/ulcer closure (wound size of 0) for two consecutive visits at least 2 weeks apart, or until the subject exited the study as treatment failure. After that, all subjects regardless of wound healing at the end of the treatment phase will be followed for 4 weeks. During the follow-up phase, standard of care will be used for subjects who have unhealed or with recurrent wounds.

At each visit, the size and changes of the target pressure ulcer are recorded by photographing. The target pressure ulcer area in the photo is calculated using Image Pro® PLUS software.

ELIGIBILITY:
1. Main inclusion criteria:

1. At least 20 years old, less than 99 (inclusive) years old, with pressure wounds located in the sacral vertebrae and greater trochanter
2. NPUAP is classified as stage 2
3. No active infection, i.e., IDSA level 1
4. Ulcer area should be ≥4 cm² and ≤25 cm² ( after necessary debridement and at time of enrollment)
5. If an artificial ostomy is not performed, the distance between the target ulcer and the anus must be greater than 5 cm to prevent contamination

2. Main exclusion criteria:

1. Those who have an allergic reaction to the ingredients of this product, including those who have been allergic to sulfa drugs, Plectranthus amboinicus, Centella asiatica or excipients
2. Acute infection caused by wound ( WBC > 12×10³/uL； or C-Reactive protein (CRP) > 30 mg/dL)
3. Liver and kidney dysfunction ( defined as [AST or ALT] > 3× the upper limit of normal; serum creatinine > 3× the upper limit of normal)
4. Pregnant or lactating women
5. Infected with human immunodeficiency virus
6. Body mass index (BMI) less than 18.5 kg/m²
7. Unable to cooperate with changing of subject's position
8. Patients with anemia (Hgb < 7.0 g/dL).
9. Unable to prevent contaminations such as feces or urinary incontinence
10. Malnutrition (Albumin< 2.5 g/dL)
11. Presence of tunneling, sinus tracts, dead spaces, etc. at the target pressure ulcer
12. In the opinion of the investigator, entering this trial may pose a threat to subject compliance.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related Adverse Events associated with Fespixon cream | 16 weeks
  Note:
  * Assessment of Safety: Safety will be assessed based on the incidence of adverse events, including overall AEs, Fespixon-related AEs, target pressure ulcer-related AEs, and SAEs.
  * During the trial, in addition to self-reported AEs, physicians will check physical examination, vital signs, and laboratory reports to determine the presence of AEs.

SECONDARY OUTCOMES:
Incidence of complete wound closure of the target ulcer area | 16 weeks
  * According to "Guidance for Industry Chronic Cutaneous Ulcer and Burn Wounds - Developing Products for Treatment" issued by the US FDA in June 2006, complete wound closure of target ulcer area is defined as "skin re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visits 2 weeks apart"
  * Time to complete wound closure of the target ulcer area was defined as "time to first visit of complete wound closure of the target ulcer area."
Time to complete wound closure of the target ulcer area | 16 weeks
  * According to "Guidance for Industry Chronic Cutaneous Ulcer and Burn Wounds - Developing Products for Treatment" issued by the US FDA in June 2006, complete wound closure of target ulcer area is defined as "skin re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visits 2 weeks apart"
  * Time to complete wound closure of the target ulcer area was defined as "time to first visit of complete wound closure of the target ulcer area."
Percentage of target ulcer wound area reduction at visit 9/ EOT (changed from V1 baseline) | 16 weeks
  Take a photo of the target ulcer and use Image-Pro® Plus software to calculate the size of the target ulcer after taking photographs.The target ulcer wound area at the Visit 9/EOT will be compared to the area of the target ulcer at the baseline visit (Visit 1) and expressed in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Hsian-Jenn Wang, Principal Investigator — Taipei Medical University WanFang Hospital; Shu-Hung Huang, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (3):
- Taiwan (3):
  - Kaohsiung Municipal Ta-Tung Hospital（Managed by Kaohsiung Medical University Chung-Ho Memorial Hospital）, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University WanFang Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
IIT study